CLINICAL TRIAL: NCT01556841
Title: A Phase II Study to Assess the Activity of TroVax® (MVA-5T4) Versus Placebo in Patients With Relapsed Asymptomatic Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: The Activity of TroVax® Versus Placebo in Relapsed Asymptomatic Ovarian Cancer
Acronym: TRIOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Oxford BioMedica (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCL/11/0119
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Randomised; Controlled; Trovax; MVA-5T4; 5T4; Immunotherapy; Relapsed; Asymptomatic; Epithelial; Ovarian; Fallopian; Peritoneal
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence | interventions — TroVax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TroVax® (Experimental): TroVax® consists of a highly attenuated VV (Modified Vaccinia Ankara, MVA) containing the human TAA 5T4 under regulatory control of a modified VV promoter, mH5.
  Interventions: Biological: TroVax®
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TroVax® — Pre-amendment 10:
  Patients will be randomised to receive either TroVax® 1 x 10↑9 TCID50/mL in 1mL (experimental arm) or matched placebo (control arm) on a 1:1 basis. A single dose will be given by intramuscular injection during the following weeks: 2, 4, 7, 10, 13, 19, 25, 31, 37, 43 and 49. No further treatment will be given beyond week 49.Treatment will be stopped early if confirmed progression or unacceptable toxicity.
  Post-amendment 10:
  Patients will be registered to receive TroVax 1 x 10↑9 TCID50/mL in 1mL only. A single dose will be given by intramuscular injection during the following weeks: 2, 4, 7, 10, 13, 19 and 25. No further treatment will be given beyond week 25.Treatment will be stopped early if confirmed progression or unacceptable toxicity.
  Arms: TroVax®
Biological: Placebo — Pre-amendment 10:
  Matched placebo will be administered as above.
  Post-amendment 10:
  TRI-70 onwards received TroVax only.
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the effectiveness of TroVax® compared to placebo in extending the time to progression in patients with asymptomatic relapsed platinum resistant ovarian, fallopian tube or primary peritoneal cancer.The trial will also look at overall survival times and quality of life.

DETAILED DESCRIPTION:
A significant number of patients with advanced ovarian cancer develop a "CA-125 relapse" without clinical symptoms and with a low volume disease on the CT scan. For this group of patients, no survival benefit has been demonstrated from early chemotherapy treatment and, on average, the time to start of chemotherapy is 5 months. Such patients could benefit from immunotherapy and the time to chemotherapy could potentially be prolonged. Multiple immunotherapy agents, such as anti-CA-125 antibodies and various vaccines, have been tested and, although there is plenty of evidence of immune response, this has not translated to a definitive clinical benefit and is not recommended in clinical practice

5T4 appears to be highly expressed in ovarian cancer and correlates with more advanced stage of disease and poorly differentiated tumours. TroVax®, the vaccine targeting 5T4, has an extensive record of safety and efficacy in humans and vaccination in patients with colorectal, renal, and prostate cancer resulted in immune cellular and humoral responses and signs of clinical benefit.

We propose a trial of TroVax® vaccination in patients with CA-125-relapsed asymptomatic ovarian cancer to assess the clinical efficacy and immunological responses as outlined in this protocol. To allow for capture of any delayed response to immunotherapy, patients who progress on RECIST 1.1 criteria and who do not experience toxicity from treatment will continue on the vaccine/placebo injection until repeat imaging at 8 weeks in order for immune-related response criteria (irRC) to be evaluated in addition to RECIST 1.1 criteria (these patients as a standard of care would not receive any other therapeutic intervention).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years with histologically or cytologically proven advanced epithelial ovarian carcinoma, fallopian tube carcinoma or primary peritoneal carcinoma
* Stage IC1 - III or Stage IVA (pleural effusion only) at diagnosis. (According to new FIGO staging effective 01/01/2014)
* Completed cytoreductive surgery during the phase of first-line therapy including removal of bulky tumour masses and adequate surgical staging including a minimum of bilateral salpingo-oophorectomy, hysterectomy and omentectomy
* Completed first line platinum-based chemotherapy OR Completed first line platinum-based chemotherapy and second line chemotherapy of any type with complete response to second line treatment according to RECIST 1.1
* Have developed relapse ≥6 months after platinum-based chemotherapy (in the case of second relapse, the disease free interval should also be ≥6 months)
* Normal CA-125 following platinum-based chemotherapy
* Have developed asymptomatic relapse as defined by:

  1. CA125 ≥ 2xULN OR
  2. Low volume radiological disease and CA125>ULN Low volume radiological disease is defined as radiologically visible disease excluding intra-hepatic (parenchymal) liver or splenic metastases, ascites or pleural effusion thought to require drainage within the next 2 months. The following are acceptable: Subcapsular liver and splenic lesions, benign lesions or cysts, any suspicious lesions that may represent metastases have to be confirmed by further imaging to be non-metastatic.
* Currently asymptomatic and does not require chemotherapy.
* Subject is assumed to be clinically immunocompetent and is free of clinically apparent/active autoimmune disease (i.e. no prior confirmed diagnosis or treatment for autoimmune disease including Systemic Lupus Erythematosis, Grave's disease, Hashimoto's thyroiditis, multiple sclerosis, and rheumatoid arthritis). Note: subjects with type I or type II diabetes mellitus can be included, as can subjects with controlled and rarely flaring rheumatoid disease (defined as recent flare within 6 months prior to randomisation/registration)
* Subject has adequate bone marrow function as defined by Haemoglobin ≥ 110 g/L, white cell count ≥ 3.0 x 10^9/L, Absolute Lymphocyte Count (ALC) ≥ 1.0 x 10^9/L, Absolute Neutrophil Count (ANC) ≥1.5 x 10^9/L , Platelet Count ≥ 100 x 10^9/L and <400 x 10^9/L, Monocytes <0.8 x 10^9/L (for patients who have undergone previous splenectomy monocyte counts can be < 1.2 x 10^9/L)
* Adequate end-organ function: plasma creatinine ≤ 2x upper limit of normal, AST and/or ALT ≤ 2x upper limit of normal, Total Bilirubin ≤ 1.5x upper limit normal
* ECOG performance status 0-1
* Life expectancy ≥6 months and willing to be available to attend clinic visits for treatment and for follow-up
* Ability to give written informed consent
* To be treated no later than 14 days from randomisation/registration

Exclusion Criteria:

* Carcino-sarcoma/MMMT
* Cancer related symptoms, or disease recurrence requiring immediate treatment
* Patients with low volume radiological disease in any of the following sites at trial entry:
* Accumulating ascites thought to require drainage within the next 2 months
* Pleural effusion thought to require drainage within the next 2 months
* Intraparenchymal Liver and/or splenic metastases
* CT scan showing bulky disease requiring chemotherapy, as judged by the investigator
* Major surgery/radiation therapy, immunotherapy or chemotherapy completed < 4 weeks prior to randomisation/registration
* Patients who are deemed as being immunosuppressed, receiving > 4 weeks parenteral or oral steroids, (nasal sprays and inhalers are permitted), or receiving immunosuppressive therapy following transplant
* Chronic (≥ 6 months) oral corticosteroid use except when prescribed as replacement therapy in the case of adrenal insufficiency. If previously used for ≥6 months then must have discontinued ≥3 months prior to randomisation/registration.
* "Currently active" second malignancy, other than non-melanoma skin cancer. Subjects are not considered to have a "currently active" malignancy if they have completed therapy ≥3 years previously and have no known evidence of residual or recurrent disease
* Concomitant use of complementary medicines/botanicals. Supplements and conventional multivitamins are acceptable.
* Evidence of significant clinical disorder or laboratory finding which in the opinion of the investigator makes it undesirable for the patient to participate in the trial. No participant should have a serious or uncontrolled intercurrent infection (including those positive for HIV, hepatitis B or C)
* Psychiatric illnesses/social situations that limit compliance with protocol requirements
* Allergy to egg proteins or history of allergic response to vaccinia vaccines
* Prior exposure to TroVax®
* Cerebral metastases (known from previous investigations or clinically detectable, surgically resected)
* Patients on active treatment as part of another clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-11; Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Progression | At 25 weeks
  Protocol-defined progression

SECONDARY OUTCOMES:
Immune-related response criteria (irRC) | 8 weeks post evidence of progression by RECIST 1.1
  irRC will be used to identify any delayed response.Patients will remain on treatment until irRc has confirmed progression (in the absence of unacceptable toxicity or the need for urgent chemotherapy).
Progression-free survival | Time from randomisation/registration to clinical intervention or confirmed evidence of progression or death, assessed for up to 2 years
Time to clinical intervention | Time from randomisation/registration to clinical intervention or death, assessed for up to 2 years
Incidence of clinical intervention | At 25 weeks from randomisation/registration
CA-125 doubling time | Assessed at treatment visits for up to 2 years from randomisation/registration.
  To investigate CA-125 doubling time as an independent prognostic factor.
Overall survival | Time between randomisation/registration and death assessed for up to 4 years
Quality of Life | For up to 2 years following randomisation/registration or until progression
  Patient reported outcome and health-related quality of life measured by standardised questionnaires (EORTC QLQ C-30, EORTC QLQ OV-28)

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Michael, MBBS, PhD, Principal Investigator — University of Surrey; Royal Surrey County Hospital NHS Foundation Trust
Locations (12):
- United Kingdom (12):
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Brighton and Sussex NHS Foundation Trust, Brighton
  - University Hospitals of Bristol NHS Foundation Trust, Bristol
  - Velindre NHS Trust, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Trust, Oxford
  - Plymouth Hospitals NHS Trust, Plymouth

REFERENCES:
- [Derived] Michael A, Wilson W, Sunshine S, Annels N, Harrop R, Blount D, Pandha H, Lord R, Ngai Y, Nicum S, Stylianou L, Gwyther S, McNeish IA, Hackshaw A, Ledermann J. A randomized phase II trial to examine modified vaccinia Ankara-5T4 vaccine in patients with relapsed asymptomatic ovarian cancer (TRIOC). Int J Gynecol Cancer. 2024 Aug 5;34(8):1225-1231. doi: 10.1136/ijgc-2023-005200. PMID 38760075
- See also: Cancer Research UK & University College London Cancer Trials Centre — http://www.ctc.ucl.ac.uk/